CLINICAL TRIAL: NCT01087489
Title: Clinical Comparison of Two Anesthetic Preparations for Intravitreal Injection
Brief Title: Comparison of Patient Comfort After Two Anesthetic Protocols for Injections Into the Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miami VA Healthcare System (U.S. Federal Agency)
Collaborators: University of Miami (Other); Bascom Palmer Eye Institute (Other)
Responsible Party: Principal Investigator, Ninel Gregori, Assistant Professor of Clinical Ophthalmology, Miami VA Healthcare System
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 00825
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Results first posted 2012-11-20 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Pain
Keywords: pain; discomfort; anesthetic drugs; topical drug administration; injections, intraocular; lidocaine; intraocular pressure; keratopathy
MeSH Terms: conditions — Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 4% lidocaine (Experimental): Eyes were anesthetized with 0.5% proparacaine and then with three cotton swabs soaked in 4% liquid lidocaine applied with moderate pressure to the site of the injection inferotemporally to the limbus. Each participant was assigned to have this prep during one of the consecutive study visits if unilateral or in one eye if patient requires bilateral injections given the same day
  Interventions: Drug: 4% lidocaine
- 3.5% ophthalmic lidocaine gel (Experimental): Eye was anesthetized with 0.5% proparacaine and then with 3.5% ophthalmic lidocaine gel applied to the surface of the eye. Each participant was randomly assigned to receive this preparation during one of two consecutive intravitreal injection (if unilateral disease) or in one eye if requiring bilateral injections given on the same day.
  Interventions: Drug: 3.5% ophthalmic lidocaine gel

INTERVENTIONS:
Drug: 4% lidocaine — The eye will be topically anesthetized with 0.5% proparacaine drops and 4% lidocaine drops and a 10% povidone-iodine scrub of the lids and lashes will be performed. A sterile speculum will be placed between the lids. Five percent povidone-iodine drops will then be applied over the ocular surface followed in three rounds by additional 5% povidone iodine and a sterile cotton swab soaked in sterile 4% lidocaine applied with gentle pressure to the area designated for injection in the infero-temporal quadrant.
  Other Names: lidocaine
  Arms: 4% lidocaine
Drug: 3.5% ophthalmic lidocaine gel — The eye will be topically anesthetized with 0.5% proparacaine drops and 5% povidone iodine will be placed over the eye. Two drops of preservative-free 3.5% lidocaine hydrochloride ophthalmic gel will be placed into inferior conjunctival sac. The patient will be asked to close the eye for 7 minutes. Next, a 10% povidone-iodine scrub of the lids and lashes will be performed. A sterile speculum will be placed between the lids. Five percent povidone-iodine drops will then be applied over the ocular surface and allowed to remain in contact with the eye for at least 2 minutes. The eye will then be rinsed with antibiotic drops.
  Other Names: Akten
  Arms: 3.5% ophthalmic lidocaine gel

SUMMARY:
Patient comfort during and after eye injections will be compared after two numbing (anesthetic) protocols, an eye preparation utilizing three cotton swabs soaked in 4% lidocaine drops versus a preparation using 3.5% lidocaine hydrochloride ophthalmic gel.

DETAILED DESCRIPTION:
The primary goal of this investigation is to determine the relative comfort of an intravitreal injection (same day and the next day) after a preparation utilizing three cotton swabs soaked in 4% lidocaine versus a preparation using 3.5% lidocaine hydrochloride ophthalmic gel. Based on the available data, the researchers contend that a preparation based on viscous 3.5% ophthalmic lidocaine gel, which coats the surface and remains in contact with the eye longer, may provide greater anesthesia and result in greater patient comfort than the topical 4% lidocaine, which is part of the standard preparation routinely utilized in the ophthalmology department currently. Secondary outcome measure is the intraocular pressure rise after the injection, and the authors will generate prospective data to study whether softening the eye with cotton swabs prior to the injection lowers post-injection pressure spike.

ELIGIBILITY:
Inclusion Criteria:

* Has required repeat Ranibizumab injections and has had at least 3 injections prior to recruitment
* Informed consent
* Age ≥ 18 years
* Clinical need for a therapeutic ranibizumab intravitreal injection regardless of the medical indication
* Able to understand and read English

Exclusion Criteria:

* Pregnancy (positive pregnancy test)
* Mental disability
* Prisoners
* Patients with fluctuating or impaired decision-making capacity
* Inability to comply with study or follow-up procedures
* Previous reaction to the same drug class

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-04; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ninel Gregori, MD, Principal Investigator — Miami VA Healthcare Systems
Locations (1):
- Miami Veterans Affairs Medical Center, Miami, Florida, United States

REFERENCES:
- [Background] Friedman SM, Margo CE. Topical gel vs subconjunctival lidocaine for intravitreous injection: a randomized clinical trial. Am J Ophthalmol. 2006 Nov;142(5):887-8. doi: 10.1016/j.ajo.2006.06.033. PMID 17056383
- [Background] Caudle LE, Williams KA, Pesudovs K. The Eye Sensation Scale: an ophthalmic pain severity measure. Optom Vis Sci. 2007 Aug;84(8):752-62. doi: 10.1097/OPX.0b013e31812f7690. PMID 17700338
- [Background] Chalam KV, Murthy RK, Agarwal S, Gupta SK, Grover S. Comparative efficacy of topical tetraVisc versus lidocaine gel in cataract surgery. BMC Ophthalmol. 2009 Aug 17;9:7. doi: 10.1186/1471-2415-9-7. PMID 19686592
- [Background] Busbee BG, Alam A, Reichel E. Lidocaine hydrochloride gel for ocular anesthesia: results of a prospective, randomized study. Ophthalmic Surg Lasers Imaging. 2008 Sep-Oct;39(5):386-90. doi: 10.3928/15428877-20080901-03. PMID 18831420
- [Background] Page MA, Fraunfelder FW. Safety, efficacy, and patient acceptability of lidocaine hydrochloride ophthalmic gel as a topical ocular anesthetic for use in ophthalmic procedures. Clin Ophthalmol. 2009;3:601-9. doi: 10.2147/opth.s4935. Epub 2009 Nov 2. PMID 19898665
- [Background] Soliman MM, Macky TA, Samir MK. Comparative clinical trial of topical anesthetic agents in cataract surgery: lidocaine 2% gel, bupivacaine 0.5% drops, and benoxinate 0.4% drops. J Cataract Refract Surg. 2004 Aug;30(8):1716-20. doi: 10.1016/j.jcrs.2003.12.034. PMID 15313296
- [Background] Bardocci A, Lofoco G, Perdicaro S, Ciucci F, Manna L. Lidocaine 2% gel versus lidocaine 4% unpreserved drops for topical anesthesia in cataract surgery: a randomized controlled trial. Ophthalmology. 2003 Jan;110(1):144-9. doi: 10.1016/s0161-6420(02)01562-2. PMID 12511360
- [Background] Cintra LP, Lucena LR, Da Silva JA, Costa RA, Scott IU, Jorge R. Comparative study of analgesic effectiveness using three different anesthetic techniques for intravitreal injection of bevacizumab. Ophthalmic Surg Lasers Imaging. 2009 Jan-Feb;40(1):13-8. doi: 10.3928/15428877-20090101-05. PMID 19205490
- [Background] Kozak I, Cheng L, Freeman WR. Lidocaine gel anesthesia for intravitreal drug administration. Retina. 2005 Dec;25(8):994-8. doi: 10.1097/00006982-200512000-00007. PMID 16340529
- [Derived] Gregori NZ, Weiss MJ, Goldhardt R, Schiffman JC, Vega E, Mattis CA, Shi W, Kelley L, Hernandez V, Feuer WJ. Ocular decompression with cotton swabs lowers intraocular pressure elevation after intravitreal injection. J Glaucoma. 2014 Oct-Nov;23(8):508-12. doi: 10.1097/IJG.0b013e318294865c. PMID 23632408
- [Derived] Gregori NZ, Weiss MJ, Goldhardt R, Schiffman JC, Vega E, Mattis CA, Shi W, Kelley L, Hernandez V, Feuer WJ. Randomized clinical trial of two anesthetic techniques for intravitreal injections: 4% liquid lidocaine on cotton swabs versus 3.5% lidocaine gel. Expert Opin Drug Deliv. 2012 Jul;9(7):735-41. doi: 10.1517/17425247.2012.685155. Epub 2012 May 3. PMID 22554019

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Miami VA Medical Center retina injection clinic; patients needing frequent intravitreal injections of ranibizumab were approached and recruited between April 2010 and March 2011
Pre-assignment Details: Patients were randomized upon recruitment and received the first anesthetic method on the day of recruitment, no wash out or transitional periods were necessary
Groups:
- Bilateral: Participants were given bilateral injections with 4% lidocaine prep in one eye and 3.5% lidocaine gel in the other.
- Unilateral: Each participant was randomly assigned to receive an intravitreal injection with 4% lidocaine prep on one visit and 3.5% lidocaine gel on the next visit.
Period: Overall Study
Arm/Group | Bilateral | Unilateral
Started | 19 | 34
Completed | 19 | 31
Not Completed | 0 | 3
Not completed — enrolled in another VA study | 0 | 1
Not completed — Death | 0 | 1
Not completed — unable to survey by telephone | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Each participant was randomly assigned to receive either anesthetic preparation during one of two consecutive intravitreal injection (if unilateral disease) or in one eye if requiring bilateral injections given on the same day.
Arm/Group | All Study Participants
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 44
Age Continuous [Mean (Standard Deviation); unit: years] | 74 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 50
Region of Enrollment [Number; unit: participants]
  United States | 53

OUTCOME MEASURES:

1. Primary Outcome: Discomfort Level and Patient Satisfaction With the Preparation Protocol and Intravitreal Injection
Description: Discomfort according to the Eye Sensation Scale: 1-none, 2- mild, 3- moderate, 4- severe, 5- extremely severe
  Patient satisfaction scale: 1=very unsatisfied, 2=unsatisfied, 3=neutral, 4=satisfied, 5= extremely satisfied
Time Frame: immediately after injection, 1- hour later, and next day
Population: all 50 patients who completed the study were included in the analysis, each patient received both anesthetic preparations prior to two consecutive (if unilateral disease) intravitreal injections on consecutive visits or in fellow eyes (if bilaterla disease) on the same day
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 4% Liquid Lidocaine Method: Each participant was randomly assigned to receive this preparation during one of two consecutive intravitreal injection (if unilateral disease) or in one eye if requiring bilateral injections given on the same day. This method involved application of 0.5% proparacaine and then 3 cotton swabs soaked in 4% liquid lidocaine applied with moderate pressure to the site of injection.
- 3.5% Ophthalmic Lidocaine Gel: Each participant was randomly assigned to receive this preparation during one of two consecutive intravitreal injection (if unilateral disease) or in one eye if requiring bilateral injections given on the same day. This method involved application of 0.5% proparacaine and then 3.5% ophthalmic lidocaine gel to the injection site.
Arm/Group | 4% Liquid Lidocaine Method | 3.5% Ophthalmic Lidocaine Gel
Number analyzed (Participants) | 50 | 50
units on a scale
  Discomfort during anesthetic preparation | 2.1 (1.1) | 2.09 (0.8)
  Discomfort during needle penetration | 1.7 (0.9) | 2.0 (0.9)
  Satisfaction with entire prep and injection | 4.3 (1.0) | 4.5 (0.8)
  Discomfort 1 h after injection | 2.4 (1.0) | 2.1 (1.1)
  Discomfort day after injection | 1.8 (0.8) | 1.6 (0.8)
  Next day satisfaction with injection | 4.3 (1.0) | 4.3 (0.9)

2. Secondary Outcome: Intraocular Pressure Change After Intravitreal Injection With Each Anesthetic Method, Results Reported in mmHg
Description: intraocular pressure (IOP) was measured immediately after the injection, and at 5, 10, and 15 minutes after the injection (until it was 30 mmHg or below). Prior to injection IOP and post-injection IOP were compared to find the IOP change after injection.
Time Frame: immediately after injection, at 5, 10, 15 minutes
Population: 48 participants were included in each arm, i.e. each participant received both methods, one eye twice if unilateral or both eyes if bilateral disease were randomily assigned to alternate prep on consecutive or same visit respectively
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | 4% Liquid Lidocaine Method | 3.5% Ophthalmic Lidocaine Gel
Number analyzed (Participants) | 48 | 48
Number analyzed (eyes) | 48 | 48
mmHg
  baseline IOP before injection | 15.5 (3.3) | 15.9 (3.0)
  IOP change after 0.05 cc injection | 25.7 (9.2) | 30.9 (9.9)

3. Secondary Outcome: Presence and Severity of Keratopathy and the Size of Subconjunctival Hemorrhage
Description: Presence of corneal staining after the injection:
  * Quadrants of fluorescein staining: 0 1 2 3 4
  * Density of staining: 0- None 1- Mild 2- Moderate 3- Severe 4- corneal abrasion
  Size of subconjunctival hemorrhage:
  in clock hours
Time Frame: within 10 minutes of the injection
Population: all eyes for which data were available were included
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | 4% Liquid Lidocaine Method | 3.5% Ophthalmic Lidocaine Gel
Number analyzed (Participants) | 49 | 49
Number analyzed (eyes) | 49 | 49
units on a scale
  Corneal fluorescein staining | 3.0 (1.0) | 2.3 (1.3)
  Density of corneal staining | 1.9 (0.7) | 1.3 (0.7)

ADVERSE EVENTS:
Arm/Group | 4% Liquid Lidocaine Method | 3.5% Ophthalmic Lidocaine Gel
Serious Adverse Events (participants affected / at risk) | 1/53 | 1/53
Other Adverse Events (participants affected / at risk) | 0/53 | 0/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4% Liquid Lidocaine Method (N=53) | 3.5% Ophthalmic Lidocaine Gel (N=53)
death (Gastrointestinal disorders) | 1 (53) | 1 (53) — death during hospitalization for general surgery

LIMITATIONS AND CAVEATS:
discomfort One hour after injection was assessed the next day via telephone and might be affected by recall bias.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No